CLINICAL TRIAL: NCT05208983
Title: SafeTy and Efficacy of Preventative CoVID Vaccines
Acronym: STOPCoV
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21-5090
Record Dates: First submitted 2022-01-24; First posted 2022-01-26 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Virus Infection; Vaccine Response
MeSH Terms: conditions — COVID-19 | interventions — mRNA Vaccines; 2019-nCoV Vaccine mRNA-1273; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dry Blood Spot specimen samples will be analyzed for vaccine induced antibodies. Remaining samples will be retained for up to 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 70 years and Older: Persons aged 70 years and over receiving a first or second dose of an approved COVID-19 vaccine and is a resident of Ontario
  Interventions: Biological: mRNA Vaccines or Viral vector-based vaccines for COVID
- 30 - 50 years of age: Persons aged 30 - 50 years receiving a first or second dose of an approved COVID-19 vaccine and a resident of Ontario
  Interventions: Biological: mRNA Vaccines or Viral vector-based vaccines for COVID

INTERVENTIONS:
Biological: mRNA Vaccines or Viral vector-based vaccines for COVID — Participants receiving an approved COVID vaccine
  Other Names: Moderna Spikevax COVID-19 vaccine; Pfizer-BioNTech Comirnaty COVID-19 vaccine; AstraZeneca Vaxzevria COVID-19 vaccine; Janssen (Johnson & Johnson) COVID-19 vaccine

SUMMARY:
The STOPCoV study is a decentralized study comparing COVID-19 vaccine specific antibody levels at 24 weeks after final vaccine dose. We plan to study the safety and immunogenicity of COVID-19 vaccine(s) in community dwelling persons 70 years and over relative to a younger group (aged 30 - 50 years).

DETAILED DESCRIPTION:
This is a prospective observational study of a cohort of individuals aged 30-50 years and a cohort of individuals aged 70 years and over receiving the COVID-19 vaccine.

Participants will complete a questionnaire to determine eligibility. Eligible participants will complete and sign an e-consent and then be provided with a participant ID, log in information and password to the database portal, and then be enrolled into the study.

Participants will complete the study assessments (baseline questionnaire, post vaccine symptom e-diary monthly, check-in questionnaire and dried blood spot specimens)

ELIGIBILITY:
Inclusion Criteria:

* Must be a resident of Ontario

Arm A:

* Individuals aged 70 and over
* Speak, read and understand English (or have a trusted individual to help with study procedures)
* Will receive a first or second dose of a COVID-19 vaccine at an Ontario vaccine distribution center. Individuals reaching the minimum age requirement by end of the recruitment calendar year are allowed to participate.

Arm B:

* Individuals between age 30-50 years
* Speak, read and understand English (or have a trusted individual to help with study procedures)
* Receive a first or second dose of a COVID-19 vaccine at an Ontario vaccine distribution center.

Exclusion Criteria:

* Not a resident of Ontario
* Individuals who are < 30 years or those 51-69 years.
* Those who are unable to complete the study protocols in English either alone or with the assistance of a trusted individual with an electronic device.
* Participants who do not receive any dose of the vaccine
* Participants who have already received both doses of the vaccine prior to enrolment.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 911 individuals ages 70 and over enrolled and 375 ages 30 - 50 enrolled
Sampling Method: Non-Probability Sample
Enrollment: 1286 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
COviD-19 vaccine specific antibody levels | 24 weeks after the final vaccination.
  The ratio-normalized levels of anti-spike and anti-RBD IgG antibodies

SECONDARY OUTCOMES:
Antibody Levels at different timepoints | 48 Weeks
  baseline, 3 weeks after first vaccine dose, prior to second dose and then at 2, 12, 36 and 48 weeks after the final vaccine dose
Safety of COVID-19 Vaccines | 48 weeks
  determine the proportion, types and severity of adverse events after the booster dose

OTHER OUTCOMES:
Breakthrough COVID Infection | 48 Weeks after the final vaccine dose
  number of persons who develop COVID post vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Walmsley, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data Sharing will be aggregate and de-identified

REFERENCES:
- See also: Study Website — http://www.stopcov.ca